CLINICAL TRIAL: NCT00074581
Title: A Randomized Trial to Evaluate the Effectiveness of Antiretroviral Therapy Plus HIV Primary Care Versus HIV Primary Care Alone to Prevent the Sexual Transmission of HIV-1 in Serodiscordant Couples
Brief Title: Preventing Sexual Transmission of HIV With Anti-HIV Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPTN 052; 10068 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2003-12-16; First posted 2003-12-17 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2016-11

CONDITIONS: HIV Infections
Keywords: HIV Infections; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Didanosine; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lamivudine; Lopinavir; lopinavir-ritonavir drug combination; Nevirapine; Stavudine; Tenofovir; lamivudine, zidovudine drug combination

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): Participants will begin ART in addition to receiving HIV primary care
  Interventions: Drug: Atazanavir; Drug: Didanosine; Drug: Efavirenz; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Stavudine; Drug: Tenofovir disoproxil fumarate; Drug: Zidovudine/Lamivudine
- 2 (Experimental): Participants will receive HIV primary care. When the CD4 count in these participants reaches 200 to 250 cells/mm3, drops below 200 cells/mm3, or develops an AIDS-defining illness, they will initiate ART.
  Note: Per LoA#5, on the Data and Safety and Monitoring Board (DSMB) recommendation, as of May 10, 2011, all HIV-infected participants in Arm 2 who have not already initiated ART will be offered ART as soon as possible.
  Interventions: Drug: Atazanavir; Drug: Didanosine; Drug: Efavirenz; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Stavudine; Drug: Tenofovir disoproxil fumarate; Drug: Zidovudine/Lamivudine

INTERVENTIONS:
Drug: Atazanavir — 300 mg taken orally once daily
  Other Names: Reyataz
Drug: Didanosine — 400 mg taken orally once daily
  Other Names: Videx
Drug: Efavirenz — 600 mg taken orally once daily
  Other Names: Sustiva
Drug: Emtricitabine/Tenofovir disoproxil fumarate — 200 mg emtricitabine/ 300 mg tenofovir disoproxil fumarate tablet taken orally once daily
  Other Names: Truvada
Drug: Lamivudine — 300 mg taken orally once daily
  Other Names: Epivir; 3TC
Drug: Lopinavir/Ritonavir — 200 mg lopinavir/ 50 mg ritonavir tablet taken orally once daily
  Other Names: Kaletra
Drug: Nevirapine — 200 mg taken orally once daily for 14 days followed by 200 mg taken orally twice daily
  Other Names: Viramune; NVP
Drug: Stavudine — Dosage depends on weight
  Other Names: Zerit; d4T
Drug: Tenofovir disoproxil fumarate — 300 mg taken orally once daily
  Other Names: Viread; TDF
Drug: Zidovudine/Lamivudine — 150 mg lamivudine/ 300 mg zidovudine tablet taken orally twice daily
  Other Names: Combivir

SUMMARY:
This study will determine whether anti-HIV drugs can prevent the sexual transmission of HIV among couples in which one partner is HIV infected and the other is not.

DETAILED DESCRIPTION:
Initiation of antiretroviral therapy (ART) in the HIV infected population has been shown to dramatically reduce the morbidity and mortality of HIV infection through sustained reduction in HIV viral replication. However, such therapy does not cure HIV infection or prevent the spread of the virus. ART may, however, make HIV infected people less contagious by lowering plasma HIV-1 RNA levels, compared with people not on ART. This study seeks to determine whether initiating ART in ART-naive, HIV infected people can prevent the sexual transmission of HIV among HIV-discordant couples, as well as to demonstrate whether quality of life changes with the initiation of ART. Both opposite and same sex couples will be recruited at study sites in Brazil, India, Malawi, Thailand, the United States, and Zimbabwe for this study.

Participating couples will be enrolled for approximately 78 months (6.5 years). Couples will be randomly assigned to one of two arms. HIV infected partners in Arm 1 will begin ART in addition to receiving HIV primary care. HIV infected partners in Arm 2 will receive HIV primary care. When the CD4 count in these participants reaches 200 to 250 cells/mm3, drops below 200 cells/mm3, or develops an AIDS-defining illness, they will initiate ART. All couples will receive HIV counseling and have their urine and blood collected at screening and enrollment, and at selected monthly, quarterly, and yearly intervals. They will be asked to periodically report information about their adherence to the ART regimen.

Note: Per LoA#5, on the Data and Safety and Monitoring Board (DSMB) recommendation, as of May 10, 2011, all HIV-infected participants in Arm 2 who have not already initiated ART will be offered ART as soon as possible.

ELIGIBILITY:
Inclusion Criteria for HIV Infected Partner:

* Positive HIV test within 60 days of study entry
* CD4 count between 350 and 550 cells/mm3 within 30 days of study entry
* If pregnant or breastfeeding, willing to be randomized to either arm of the study

Inclusion Criteria for HIV Uninfected Partner:

* Negative HIV test within 14 days of study entry

Inclusion Criteria for Both Partners:

* Plans to maintain sexual relationship with partner
* Reports having sex (vaginal or anal) with partner at least three times in the last 3 months
* Willing to disclose HIV test results to partner
* Plans to stay in the area and does not have a job or other obligations that may require long absences during the duration of the study

Exclusion Criteria for HIV Infected Partner:

* Current or previous use of any ART. Participants who previously took a short-term course of ART for prevention of mother-to-child transmission of HIV are not excluded.
* Documented or suspected acute hepatitis within 30 days of study entry, if the infected partner's starting regimen in the study contains nevirapine or atazanavir
* Current or previous AIDS-defining illness or opportunistic infection
* Documented or suspected acute hepatitis within 30 days prior to study entry
* Acute therapy of serious medical illnesses within 14 days prior to study entry
* Radiation therapy or systemic chemotherapy within 45 days prior to study entry
* Immunomodulatory or investigational therapy within 30 days prior to study entry
* Active drug or alcohol dependence that, in the opinion of the investigator, would interfere with the study
* Vomiting or inability to swallow medications
* Require certain medications
* Allergy or sensitivity to any of the study drugs

Exclusion Criteria for Both Partners:

* History of injection drug use within 5 years of study entry
* Previous and/or current participation in an HIV vaccine study
* Currently detained in jail or for treatment of a psychiatric or physical illness
* Any condition that, in the opinion of the study staff, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives
* Certain abnormal laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3526 (Actual)
Dates: Start 2005-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron S. Cohen, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (17):
- Fenway Community Health Ctr. CRS, Boston, Massachusetts, United States
- Gaborone CRS, Gaborone, Botswana
- Brazil (4):
  - Hospital Geral de Nova Iguaçu CRS (HGNI CRS), Nova Iguaçu, Rio de Janeiro
  - Hospital Nossa Senhora da Conceicao CRS, Port Alegre, Rio Grande do Sul
  - HSE-Hospital dos Servidores do Estado CRS, Rio de Janeiro
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
- India (4):
  - NARI Clinic at Gadikhana Dr. Kotnis Municipal Dispensary CRS, Pune, Maharashtra
  - NARI Clinic at NIV CRS, Pune, Maharashtra
  - NARI Pune CRS, Pune, Maharashtra
  - Chennai Antiviral Research and Treatment (CART) CRS, Chennai, Tamil Nadu
- Kisumu Crs, Kisumu, Nyanza, Kenya
- Malawi (2):
  - Blantyre CRS, Blantyre
  - Malawi CRS, Lilongwe
- South Africa (2):
  - Soweto HPTN CRS, Johannesburg, Gauteng
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS), Johannesburg, Gauteng
- CMU HIV Prevention CRS, Chiang Mai, Thailand
- Parirenyatwa CRS, Harare, Zimbabwe

REFERENCES:
- [Background] Chan DJ. Fatal attraction: sex, sexually transmitted infections and HIV-1. Int J STD AIDS. 2006 Oct;17(10):643-51. doi: 10.1258/095646206780071018. PMID 17059632
- [Background] Chan DJ. Factors affecting sexual transmission of HIV-1: current evidence and implications for prevention. Curr HIV Res. 2005 Jul;3(3):223-41. doi: 10.2174/1570162054368075. PMID 16022655
- [Background] Davis CW, Doms RW. HIV transmission: closing all the doors. J Exp Med. 2004 Apr 19;199(8):1037-40. doi: 10.1084/jem.20040426. Epub 2004 Apr 12. No abstract available. PMID 15078894
- [Background] Gupta K, Klasse PJ. How do viral and host factors modulate the sexual transmission of HIV? Can transmission be blocked? PLoS Med. 2006 Feb;3(2):e79. doi: 10.1371/journal.pmed.0030079. Epub 2006 Feb 28. PMID 16492075
- [Derived] Odero I, Ondeng'e K, Mudhune V, Okola P, Oruko J, Otieno G, Akelo V, Gust DA. Participant satisfaction with clinical trial experience and post-trial transitioning to HIV care in Kenya. Int J STD AIDS. 2019 Jan;30(1):12-19. doi: 10.1177/0956462418791946. Epub 2018 Aug 29. PMID 30157702
- [Derived] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Cottle L, Zhang XC, Makhema J, Mills LA, Panchia R, Faesen S, Eron J, Gallant J, Havlir D, Swindells S, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano DD, Essex M, Hudelson SE, Redd AD, Fleming TR; HPTN 052 Study Team. Antiretroviral Therapy for the Prevention of HIV-1 Transmission. N Engl J Med. 2016 Sep 1;375(9):830-9. doi: 10.1056/NEJMoa1600693. Epub 2016 Jul 18. PMID 27424812
- [Derived] Grinsztejn B, Hosseinipour MC, Ribaudo HJ, Swindells S, Eron J, Chen YQ, Wang L, Ou SS, Anderson M, McCauley M, Gamble T, Kumarasamy N, Hakim JG, Kumwenda J, Pilotto JH, Godbole SV, Chariyalertsak S, de Melo MG, Mayer KH, Eshleman SH, Piwowar-Manning E, Makhema J, Mills LA, Panchia R, Sanne I, Gallant J, Hoffman I, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Havlir D, Cohen MS; HPTN 052-ACTG Study Team. Effects of early versus delayed initiation of antiretroviral treatment on clinical outcomes of HIV-1 infection: results from the phase 3 HPTN 052 randomised controlled trial. Lancet Infect Dis. 2014 Apr;14(4):281-90. doi: 10.1016/S1473-3099(13)70692-3. Epub 2014 Mar 4. PMID 24602844
- [Derived] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103

RESULTS

PARTICIPANT FLOW:
Groups:
- Early-ART: Participants will begin ART in addition to receiving HIV primary care
  Atazanavir: 300 mg taken orally once daily
  Didanosine: 400 mg taken orally once daily
  Efavirenz: 600 mg taken orally once daily
  Emtricitabine/Tenofovir disoproxil fumarate: 200 mg emtricitabine/ 300 mg tenofovir disoproxil fumarate tablet taken orally once daily
  Lamivudine: 300 mg taken orally once daily
  Lopinavir/Ritonavir: 200 mg lopinavir/ 50 mg ritonavir tablet taken orally once daily
  Nevirapine: 200 mg taken orally once daily for 14 days followed by 200 mg taken orally twice daily
  Stavudine: Dosage depends on weight
  Tenofovir disoproxil fumarate: 300 mg taken orally once daily
  Zidovudine/Lamivudine: 150 mg lamivudine/ 300 mg zidovudine tablet taken orally twice daily
  Note: Sites could also use locally supplied, FDA-approved drugs if they could be purchased with nonstudy funds. For participants with virologic failure, specified second-line treatment regimens were provided.
- Delayed-ART: Participants will receive HIV primary care. When the CD4 count in these participants reaches 200 to 250 cells/mm3, drops below 200 cells/mm3, or develops an AIDS-defining illness, they will initiate ART.
  (Same drug regimen as that described in the early-ART arm)
  Note: Per LoA#5, on the Data and Safety and Monitoring Board (DSMB) recommendation, as of May 10, 2011, all HIV-infected participants in Arm 2 who have not already initiated ART will be offered ART as soon as possible.
Period: Overall Study
Arm/Group | Early-ART | Delayed-ART
Started | 1789 (886 HIV-infected index cases and 903 HIV-uninfected partners) | 1767 (877 HIV-infected index cases and 890 HIV-uninfected partners)
Completed | 1545 | 1541
Not Completed | 244 | 226
Not completed — Death | 15 | 16
Not completed — Withdrawal by Subject | 50 | 49
Not completed — Unable to adhere to visit schedule | 13 | 14
Not completed — Relocated | 14 | 9
Not completed — Were withdrawn by investigator | 5 | 2
Not completed — Lost to Follow-up | 16 | 11
Not completed — Ended relationship w. index participant | 117 | 106
Not completed — Other | 14 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-ART | Delayed-ART | Total
Number analyzed (Participants) | 1789 | 1767 | 3556
Age, Customized [Number; unit: participants]
  18-25 yr | 300 | 335 | 635
  26-40 yr | 1101 | 1079 | 2180
  >40 yr | 388 | 353 | 741
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 877 | 860 | 1737
  Male | 912 | 907 | 1819
Region [Number; unit: participants]
  North or South America | 293 | 279 | 572
  Asia | 535 | 528 | 1063
  Africa | 961 | 960 | 1921

OUTCOME MEASURES:

1. Primary Outcome: Linked Partner HIV Infection Rates in Early-ART and Delayed-ART Arms
Description: incident HIV infections occurring in the partners (HIV-negative at enrollment) of randomized HIV-infected index (HIV-positive at enrollment) cases are assessed, by arm. Only acquisition from the index partner were included in the primary analysis, therefore, each endpoint was required to be confirmed (by genotyping) such that the viral envelop sequence in the index case matched that of the partner.
Time Frame: Throughout study
Measure: Number (95% Confidence Interval); unit: event rate per 100 person-yr
Units Other Than Participants: Person Years
Arm/Group | Early-ART | Delayed-ART
Number analyzed (Participants) | 903 | 890
Number analyzed (Person Years) | 4325 | 4185
event rate per 100 person-yr | 0.07 [0.01 to 0.20] | 1.03 [0.74 to 1.38]
Statistical Analysis 1: Comparison: Early-ART vs Delayed-ART; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.07, 95% CI 2-sided [0.02 to 0.22] — The hazard ratio estimate presented (0.07) is a comparison of the early-ART arm (numerator) to the delayed-ART arm (denominator), thus indicating a 93% lower risk of infection among all linked partner infections, during the entire study

2. Primary Outcome: All Partner HIV Infection Rates in Early-ART and Delayed-ART Arms
Description: All Incident HIV infections occurring in the partners (HIV-negative at enrollment) of randomized HIV-infected index (HIV-positive at enrollment) cases are assessed, by arm.
Time Frame: Throughout study
Population: Population includes all partners (HIV-negative at enrollment) of randomized HIV-infected index (HIV-positive at enrollment) cases, by arm.
Measure: Number (95% Confidence Interval); unit: event rate per 100 person-yr
Arm/Group | Early-ART | Delayed-ART
Number analyzed (Participants) | 903 | 890
event rate per 100 person-yr | 0.44 [0.26 to 0.69] | 1.41 [1.07 to 1.82]
Statistical Analysis 1: Comparison: Early-ART vs Delayed-ART; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.19 to 0.53] — The hazard ratio estimate presented (0.31) is a comparison of the early-ART arm (numerator) to the delayed-ART arm (denominator), thus indicating a 69% lower risk of infection among all partner infections, during the entire study

ADVERSE EVENTS:
Description: Only index participants were monitored for adverse events since they (and not partners) were receiving treatment drugs.
Arm/Group | Early-ART | Delayed-ART
Serious Adverse Events (participants affected / at risk) | 526/886 | 522/877
Other Adverse Events (participants affected / at risk) | 0/886 | 0/877
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early-ART (N=886) | Delayed-ART (N=877)
Anaemia (Blood and lymphatic system disorders) | 15 | 19
Anaemia of pregnancy (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 — General disorders as well as administration site conditions
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 62 | 66
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1
Congenital anomaly in offspring (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 6
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 7
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 6 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 7 | 5
Fatigue (General disorders) | 3 | 2
Hyperthermia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Injection site pain (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Polyp (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 5
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 4 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 2
Hepatotoxicity (Hepatobiliary disorders) | 6 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 37 | 14
Liver disorder (Hepatobiliary disorders) | 1 | 5
Anaphylactic reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 3
Abortion infected (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess bacterial (Infections and infestations) | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 4
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 4
Cerebral malaria (Infections and infestations) | 1 | 1
Dengue fever (Infections and infestations) | 1 | 4
Diarrhoea infectious (Infections and infestations) | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 2
Dysentery (Infections and infestations) | 1 | 4
Enteritis infectious (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Extrapulmonary tuberculosis (Infections and infestations) | 1 | 6
Furuncle (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 12 | 19
Gastrointestinal infection (Infections and infestations) | 0 | 2
H1N1 influenza (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 5
Herpes zoster oticus (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 2
Joint abscess (Infections and infestations) | 0 | 1
Leptospirosis (Infections and infestations) | 4 | 2
Liver abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lymph node tuberculosis (Infections and infestations) | 0 | 2
Malaria (Infections and infestations) | 23 | 20
Measles (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 4 | 2
Meningitis bacterial (Infections and infestations) | 1 | 1
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 2
Meningococcal sepsis (Infections and infestations) | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1
Nasal abscess (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 8 | 6
Pharyngitis (Infections and infestations) | 0 | 3
Pharyngitis bacterial (Infections and infestations) | 1 | 1
Plasmodium falciparum infection (Infections and infestations) | 2 | 0
Plasmodium malariae infection (Infections and infestations) | 3 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 16 | 11
Pneumonia bacterial (Infections and infestations) | 7 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 4 | 7
Pyelonephritis (Infections and infestations) | 2 | 2
Pyelonephritis acute (Infections and infestations) | 2 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Secondary syphilis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 2 | 3
Tonsillitis bacterial (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 2 | 0
Tracheobronchitis (Infections and infestations) | 2 | 0
Tuberculosis (Infections and infestations) | 1 | 1
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 1
Typhoid fever (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 3
Viral infection (Infections and infestations) | 0 | 4
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 0 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Hair injury (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 3 | 0
Alanine aminotransferase increased (Investigations) | 20 | 19
Aspartate aminotransferase increased (Investigations) | 32 | 29
Blood albumin decreased (Investigations) | 6 | 9
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bicarbonate decreased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 68 | 42
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 7
Blood glucose increased (Investigations) | 1 | 1
Blood phosphorus decreased (Investigations) | 73 | 86
Blood phosphorus increased (Investigations) | 0 | 2
Blood potassium decreased (Investigations) | 3 | 1
Blood potassium increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 8 | 8
Blood sodium increased (Investigations) | 3 | 2
Blood triglycerides increased (Investigations) | 2 | 2
Haemoglobin decreased (Investigations) | 15 | 18
Hepatic enzyme increased (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 0 | 2
Low density lipoprotein increased (Investigations) | 2 | 2
Neutrophil count decreased (Investigations) | 64 | 80
Platelet count decreased (Investigations) | 8 | 19
Transaminases increased (Investigations) | 6 | 9
White blood cell count decreased (Investigations) | 1 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 75 | 54
Decreased appetite (Metabolism and nutrition disorders) | 2 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 5
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 42 | 43
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Choriocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Ataxia (Nervous system disorders) | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Diplegia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 14 | 8
Dizziness postural (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Febrile convulsion (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 6
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 3 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tonic convulsion (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 6 | 7
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2 | 3
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 9 | 16
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 4
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 3 | 2
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 4 | 1
Acute psychosis (Psychiatric disorders) | 1 | 1
Acute stress disorder (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Brief psychotic disorder, with postpartum onset (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 5 | 3
Confusional state (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 4
Drug abuse (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 1
Homicidal ideation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Intentional self-injury (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 4 | 3
Mental disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 3 | 0
Suicidal ideation (Psychiatric disorders) | 12 | 5
Suicide attempt (Psychiatric disorders) | 8 | 5
Violence-related symptom (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 4
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 2
Urogenital fistula (Renal and urinary disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 3 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 3 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 3 | 0
Menorrhagia (Reproductive system and breast disorders) | 4 | 5
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 3 | 2
Ovarian cyst (Reproductive system and breast disorders) | 2 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Victim of homicide (Social circumstances) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 7 | 5
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 8 | 9
Systolic hypertension (Vascular disorders) | 0 | 1
Thromboangiitis obliterans (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study abstracts and publications are subject to HPTN Publication and Public Information Policies and Clinical Trial Agreements between NIAID (DAIDS) and company collaborators. The publication or other disclosure can be delayed for up to thirty additional business days for manuscripts and five business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.